CLINICAL TRIAL: NCT05662800
Title: Development of Peanut, Sesame, and Tree Nut Allergy in Polish Children at High Risk of Food Allergy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Nutricia Foundation (Other); Thermo Fisher Scientific, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: RG 2/2021
Record Dates: First submitted 2022-12-05; First posted 2022-12-23 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Atopic Dermatitis; Food Allergy; Peanut Allergy; Tree Nut Allergy
Keywords: atopic dermatitis; peanuts; tree nuts; sesame; food allergy; children
MeSH Terms: conditions — Dermatitis, Atopic; Food Hypersensitivity; Peanut Hypersensitivity; Nut Hypersensitivity; SeSAME syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Assessment of peanut, tree nuts and sesame allergy — Children will undergo skin prick testing with the following allergens: commercial extracts for peanut, hazelnut, almond, cashew, pistachio, walnut, macadamia, sesame, Timothy grass, and birch pollen; positive and negative control; peanut butter and tahini (sesame) paste.
  Specific IgE levels will be quantified to all the above-listed tree nuts, peanuts, sesame seed and peanut components (Ara h 1, Ara h 2, Ara h 3, Ara h 6, Ara h 8, Ara h 9).
  Children will undertake cumulative or incremental oral food challenge with peanut, sesame and tree nuts, depending on the risk assessment based on patient's medical history and results of diagnostic tests.

SUMMARY:
The aim of the study is to assess the prevalence of peanut, tree nuts, and sesame allergy in Polish children at high risk of food allergy. Additionally, the timing of the development of peanut, tree nuts and sesame allergy in the first three years of life in a high-risk population will be assessed.

DETAILED DESCRIPTION:
Introduction: Peanut allergy (PA) has become a health concern world-wide for several decades. Sesame allergy, although less prevalent, is also causing growing concern. Peanut, tree nuts, and sesame allergy co-exist in 60% of children. Although the majority of PA cases come from the general population, there are well-established risk factors for this allergy, such as eczema and egg allergy. In the Learning Early About Peanut (LEAP) Study, early introduction of peanut into the diet of children with moderate-to-severe eczema or egg allergy was proven to be effective in PA prevention. This strategy has now been adopted by national allergy societies in the USA and Australia as part of the weaning guidance for the high-risk populations.However, it is not known whether early introduction of peanut is also justified in other populations where peanut consumption has traditionally been lower. Getting insight into the prevalence of nut and sesame allergy in the cohort of infants and toddlers in Central Europe is needed to guide early dietary intervention strategies.

Methods: 240 children with eczema or egg allergy will undertake extensive assessment of peanut, tree nuts (hazelnut, almond, cashew, pistachio, walnut, macadamia) and sesame allergy status through consumption history, skin testing, specific immunoglobulin E measurement (sIgE) and oral food challenges (OFCs).

ELIGIBILITY:
Inclusion Criteria:

* moderate or severe eczema and/or egg allergy,
* at least one complementary food already introduced,
* signed informed consent.

Assessment of eczema severity: Eczema severity will be assessed based on the objective SCORing Atopic Dermatitis (SCORAD), use of topical steroids, calcineurin inhibitors or systemic treatment as well as history of hospital admission.

Definition of egg allergy: Participants with a documented IgE-mediated egg allergy will be identified by a convincing history of a reaction in the presence of a positive skin prick test (SPT) (wheal diameter of 3 mm or greater with egg white extract) or an SPT ≥ 5mm with no history of a reaction.

Exclusion Criteria:

* inability to withdraw antihistamines for at least 5 days prior to testing,
* use of prohibited medication such as beta-blockers, angiotensin-converting-enzyme inhibitors (ACE-I) and biological treatments affecting the immunological response,
* uncontrolled asthma or eczema which does not warrant readiness for a food challenge within the study time frame,
* chronic urticaria,
* chronic systemic diseases.

Ages: 4 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The children will be recruited using mailing to general paediatric, allergy, and dermatology practices and directly to two allergy centers (Warsaw and Bydgoszcz).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
The prevalence of peanut, tree nut and sesame allergy in Polish children with high risk of food allergy | 1-2 days
  Based on data related to allergen consumption, SPT, and OFC, patients will be classified as allergic to peanuts and sesame or non-allergic. Based on the results of SPT, sIgE, and OFCs are performed in exceptional situations, patients will be classified as allergic, non-allergic, or likely not allergic to selected tree nuts.

OTHER OUTCOMES:
The timing of the development of peanut, tree nuts and sesame allergy in the first three years of life in a high-risk population | 2 years
  Assessment of the prevalence of peanuts, tree nuts and sesame allergy (based on data related to allergen consumption, SPT, sIgE and OFC; as described in Outcome 1) will be performed in the investigated group with ensured equal representation of age. The study will aim to recruit 20% of children aged 4 to 6 months, 15% aged 7 to 9 months, 15% aged 10 to 12 months, 15% aged 13 to 18 months, 15% aged 19 to 24 months and 20% in the third year of life.

CONTACTS AND LOCATIONS:
Overall Officials: Marek Kulus, MD, Prof., Principal Investigator — Medical University of Warsaw
Locations (2):
- Poland (2):
  - Department of Pediatric Pneumonology and Allergy, Medical University of Warsaw, Warsaw, Masovian Voivodeship
  - Department of Pediatrics, Allergology and Gastroenterology, Collegium Medicum in Bydgoszcz, Nicolaus Copernicus University, Bydgoszcz

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or generated during this study will be made available after the publication of results, no later than 3 years from the completion of data analysis.
Supporting Information: CSR
Time Frame: Up to 3 years after completion of data analysis.
Access Criteria: The datasets will be made available from the contact author upon reasonable request.

REFERENCES:
- [Background] Brough HA, Caubet JC, Mazon A, Haddad D, Bergmann MM, Wassenberg J, Panetta V, Gourgey R, Radulovic S, Nieto M, Santos AF, Nieto A, Lack G, Eigenmann PA. Defining challenge-proven coexistent nut and sesame seed allergy: A prospective multicenter European study. J Allergy Clin Immunol. 2020 Apr;145(4):1231-1239. doi: 10.1016/j.jaci.2019.09.036. Epub 2019 Dec 20. PMID 31866098
- [Background] Du Toit G, Roberts G, Sayre PH, Bahnson HT, Radulovic S, Santos AF, Brough HA, Phippard D, Basting M, Feeney M, Turcanu V, Sever ML, Gomez Lorenzo M, Plaut M, Lack G; LEAP Study Team. Randomized trial of peanut consumption in infants at risk for peanut allergy. N Engl J Med. 2015 Feb 26;372(9):803-13. doi: 10.1056/NEJMoa1414850. Epub 2015 Feb 23. PMID 25705822
- [Background] Perkin MR, Logan K, Tseng A, Raji B, Ayis S, Peacock J, Brough H, Marrs T, Radulovic S, Craven J, Flohr C, Lack G; EAT Study Team. Randomized Trial of Introduction of Allergenic Foods in Breast-Fed Infants. N Engl J Med. 2016 May 5;374(18):1733-43. doi: 10.1056/NEJMoa1514210. Epub 2016 Mar 4. PMID 26943128
- [Background] Du Toit G, Katz Y, Sasieni P, Mesher D, Maleki SJ, Fisher HR, Fox AT, Turcanu V, Amir T, Zadik-Mnuhin G, Cohen A, Livne I, Lack G. Early consumption of peanuts in infancy is associated with a low prevalence of peanut allergy. J Allergy Clin Immunol. 2008 Nov;122(5):984-91. doi: 10.1016/j.jaci.2008.08.039. PMID 19000582
- [Background] Togias A, Cooper SF, Acebal ML, Assa'ad A, Baker JR Jr, Beck LA, Block J, Byrd-Bredbenner C, Chan ES, Eichenfield LF, Fleischer DM, Fuchs GJ 3rd, Furuta GT, Greenhawt MJ, Gupta RS, Habich M, Jones SM, Keaton K, Muraro A, Plaut M, Rosenwasser LJ, Rotrosen D, Sampson HA, Schneider LC, Sicherer SH, Sidbury R, Spergel J, Stukus DR, Venter C, Boyce JA. Addendum guidelines for the prevention of peanut allergy in the United States: Report of the National Institute of Allergy and Infectious Diseases-sponsored expert panel. J Allergy Clin Immunol. 2017 Jan;139(1):29-44. doi: 10.1016/j.jaci.2016.10.010. PMID 28065278
- [Derived] Ryczaj K, Szczukocka-Zych A, Wawszczak M, Gawryjolek J, Krogulska A, Krawiec M, Horvath A, Szajewska H, Santos A, Bahnson HT, Kulus M. Development of peanut, sesame and tree nut allergy in Polish children at high risk of food allergy: a protocol for a cross-sectional study. BMJ Open. 2023 Nov 16;13(11):e074168. doi: 10.1136/bmjopen-2023-074168. PMID 37973545